CLINICAL TRIAL: NCT02751944
Title: Evaluation of the Effects of NEM® Brand Eggshell Membrane Versus Placebo on Exercise-induced Joint Pain, Stiffness, & Cartilage Turnover in Healthy, Post-menopausal Women
Brief Title: NEM® Versus Placebo on Exercise-induced Joint Pain, Stiffness, & Cartilage Turnover In Healthy, Post-Menopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ESM Technologies, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: ESM-CLN#2015T02
Record Dates: First submitted 2016-04-22; First posted 2016-04-26 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Exercise-induced Joint Pain Stiffness and Cartilage Turnover
Keywords: exercise-induced; joint pain; joint stiffness; post-menopausal; women; cartilage turnover; CTX-II
MeSH Terms: conditions — Arthralgia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NEM Treatment (Experimental): NEM, 500 mg, once daily, orally for 2 weeks
  Interventions: Dietary Supplement: NEM
- Placebo (Placebo Comparator): Placebo, 500 mg, once daily, orally for 2 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: NEM — Dietary supplement for the support of joint health.
  Other Names: Natural Eggshell Membrane
  Arms: NEM Treatment
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study is intended to evaluate the effect of the dietary supplement NEM® brand eggshell membrane versus placebo in reducing exercise-induced joint pain & stiffness & cartilage turnover in healthy post-menopausal women. Half of the study participants will receive NEM, once daily, orally while the other half of the study participants will receive placebo, once daily, orally.

DETAILED DESCRIPTION:
Moderate exercise can induce discomfort in joints when done infrequently or when done too intensely or for too long a period. This discomfort is often realized as either pain or stiffness in the joint that was the focus of the exercise. For example, one's knees will hurt after jogging for several miles, particularly if jogging for the first time. This study is intended to evaluate whether NEM® brand eggshell membrane can alleviate joint pain or stiffness, either directly following exercise or 12 hours post-exercise versus placebo. The study will also evaluate NEM's effect, if any, on cartilage turnover via the cartilage degradation biomarker c-terminal cross-linked telopeptide of type II collagen (CTX-II). Participants will perform a minimum of 50 steps per leg utilizing an aerobics step at the clinical site. They will follow this exercise regimen on alternating days for 2 weeks. Changes in pain & stiffness (immediate & 12-hour) will be compared to both baseline and to the placebo group. Blood & Urine samples will also be collected at baseline and at the end of Week 1 & Week 2. The change in CTX-II will be compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be female, 40-75 years of age.
2. Subject must have been amenorrheic (post-menopausal) for at least 12 months prior to baseline evaluation, either naturally or surgically.
3. Subject must not have been diagnosed with a joint or connective tissue (JCT) disease (i.e. osteoarthritis, rheumatoid arthritis, spondyloarthritis, bursitis, gout, systemic lupus erythematosus, fibromyalgia, etc.) affecting the hip, knee, or ankle by a licensed physician prior to enrollment evaluation.
4. Subjects must have a resting pain/discomfort score of ≤ 3 on the 10 point Likert scale in the knee with the most severe pain/discomfort.
5. Subject must be willing and healthy enough to perform moderate exercise.
6. Subject must be available for and willing to attend all evaluation visits.
7. Subject must be able and willing to give informed consent.
8. Subjects must be willing to use only acetaminophen as rescue pain medication, if needed.
9. Subjects participating in prior studies evaluating eggshell membrane can participate in the current study so long as they are not currently taking an eggshell membrane supplement and have not done so for 60 days prior to screening.

Exclusion Criteria:

1. Subject is currently receiving therapy with remission-inducing drugs (i.e. methotrexate, tumor necrosis factor (TNF) biologics, etc.), immunosuppressive drugs (i.e. corticosteroids, transplantation medications, etc.).
2. Subject has been diagnosed with any clinically significant confounding inflammatory disease or condition that would interfere with the study evaluation, as judged by the clinical investigator (i.e. pseudo gout, Paget's disease, chronic pain syndrome, active rheumatic fever, etc.).
3. Subject has a known allergy to eggs or egg products. If any subject becomes sensitive during the study, they will immediately be excluded from continuing in the study.

   a. Such sensitivity may be realized as a reaction to inoculations wherein the inoculate is derived from or contains egg components (i.e., influenza vaccine).
4. Subject suffers from clinically significant cardiac, pulmonary, or other complications that would prevent them from performing moderate exercise or could pose a risk to the subject's health, as judged by the clinical investigator.
5. Subject participates in activities involving intensive use of the lower extremities (i.e. running / jogging, sports, bicycling, dancing, etc.) 2 or more days per week or participates in activities that involve moderate use of the lower extremities (i.e. walking, golfing, yoga, etc.) 3 or more days per week.
6. Subject body weight is greater than 275 pounds (125 kg).
7. Subject is currently taking or is unwilling to forgo the use of prescription, over-the-counter (OTC) treatments, and/or dietary supplements affecting joint health within 30 days prior to baseline evaluation and for the duration of the study. Prohibited medications include: NSAIDs, analgesics (other than acetaminophen), opioids, anti-depressants prescribed for painful conditions (i.e. fibromyalgia) & joint supplements. Examples of these types of medications are: aspirin, ibuprofen, naproxen, oxycodone, propoxyphene, diclofenac, celecoxib, amitriptyline, duloxetine, glucosamine, chondroitin, MSM, white willow bark, turmeric or curcumin, Boswellia, fish oil, etc.

   a. Washout Periods: Subjects are eligible to participate in the study following a 7-day washout period for opioids, a 14-day washout period for analgesics & NSAIDs, and a 90-day washout period for steroids, anti-depressants, or JCT dietary supplements (i.e. glucosamine, chondroitin, methylsulfonylmethane (MSM), etc.) Acetaminophen must not have been taken within 24 hours of baseline evaluation.
8. Subject is involved in any other research study involving an investigational product (drug, device or biologic) or a new application of an approved product, within 30 days of baseline evaluation.
9. Pregnant and breastfeeding women.
10. Subject has a history or positive test result of HIV, hepatitis B or hepatitis C.

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-12; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Exercise-induced Cartilage Turnover via CTX-II Biomarker | 2 weeks
  To evaluate the efficacy of NEM® versus placebo at reducing exercise-induced cartilage turnover in healthy, post-menopausal women by evaluating the change in urinary CTX-II levels.

SECONDARY OUTCOMES:
Exercise-induced Joint Pain via questionnaire | 2 weeks
  To evaluate the efficacy of NEM® versus placebo at reducing exercise-induced knee discomfort (pain/aching) based upon perceived pain rated on a 10 point Likert scale.
Exercise-induced Joint Stiffness via questionnaire | 2 weeks
  To evaluate the efficacy of NEM® versus placebo at reducing exercise-induced knee stiffness based upon perceived stiffness rated on a 10 point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Morrison, D.O., Principal Investigator — QPS-Biokinetic; Kevin J Ruff, Ph.D., MBA, Study Director — ESM Technologies, LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ruff KJ, Morrison D, Duncan SA, Back M, Aydogan C, Theodosakis J. Beneficial effects of natural eggshell membrane versus placebo in exercise-induced joint pain, stiffness, and cartilage turnover in healthy, postmenopausal women. Clin Interv Aging. 2018 Feb 19;13:285-295. doi: 10.2147/CIA.S153782. eCollection 2018. PMID 29497287
- See also: Published in Clinical Interventions in Aging — https://doi.org/10.2147/CIA.S153782